CLINICAL TRIAL: NCT01190995
Title: A Randomised Controlled Trial to Evaluate the Role of Repeated Painful Procedures in Preterm Neonates on Short Term Neurobehavioural Outcome
Brief Title: Role of Repeated Painful Procedures in Preterm Neonates on Short Term Neurobehavioural Outcome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, DR. VIKRAM DATTA, Professor, Lady Hardinge Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: Pain and Neurobehaviour
Record Dates: First submitted 2010-08-27; First posted 2010-08-30 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Pain
Keywords: Pain; Neonate; Procedure; Neurobehavioural outcome
MeSH Terms: conditions — Pain | interventions — Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sucrose (Experimental): The enrolled neonates will be administered a sterile solution of 24 % sucrose orally for a period of 7 days from enrollment The patient will be enrolled into the study only after an informed written consent has been obtained from either of the parent/caregiver. At the beginning of each potentially painful procedure namely, venepuncture, venous and arterial cannulation, heel lance,orogastric tube insertion, suprapubic aspiration of urine and any other skin breaking procedure,0.5ml of solution marked with patients serial number will be administered by a prefilled syringe to the patient on the anterior aspect of the tongue , avoiding spillage , by the personnel carrying out the procedure.
  Interventions: Drug: 24% Sucrose; Drug: Placebo
- Placebo (Placebo Comparator): The enrolled neonates will be administered double distilled water orally for a period of 7 days from enrollment. At the beginning of each potentially painful procedure namely, venepuncture, venous and arterial cannulation, heel lance,orogastric tube insertion, suprapubic aspiration of urine and any other skin breaking procedure,0.5ml of solution marked with patients serial number will be administered by a prefilled syringe to the patient on the anterior aspect of the tongue , avoiding spillage , by the personnel carrying out the procedure
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 24% Sucrose — The enrolled neonates will be administered either a sterile solution of 24 % sucrose or double distilled water orally for a period of 7 days from enrollment. At the beginning of each potentially painful procedure namely, venepuncture, venous and arterial cannulation, heel lance,orogastric tube insertion, suprapubic aspiration of urine and any other skin breaking procedure,0.5ml of solution marked with patients serial number will be administered by a prefilled syringe to the patient on the anterior aspect of the tongue , avoiding spillage , by the personnel carrying out the procedure
  Other Names: Sucrose
  Arms: Sucrose
Drug: Placebo — The patient will be enrolled into the study only after an informed written consent has been obtained from either of the parent/caregiver. At the beginning of each potentially painful procedure namely, venepuncture, venous and arterial cannulation, heel lance,orogastric tube insertion, suprapubic aspiration of urine and any other skin breaking procedure,0.5ml of solution marked with patients serial number will be administered by a prefilled syringe to the patient on the anterior aspect of the tongue , avoiding spillage , by the personnel carrying out the procedure
  Other Names: Distilled Water

SUMMARY:
Procedural pain in neonates is recently acknowledged entity and many studies on the use of pharmacological as well as non pharmacological interventions for alleviation of this pain have been done. Of these, sucrose with or without non nutritive sucking has been the most widely studied and accepted form of pain relief. Its analgesic effect is thought to be mediated by endogenous opioid pathways activated by sweet taste (orogustatory effect).

Although, guidelines based on systematic reviews and meta-analysis for pain management recommend the use of sucrose solutions for pain relief during procedures, the use of repeated doses of sucrose with preterm neonates requires further investigation.

Pain may have profound consequences for preterm neonates during a critical time of brain development. Data derived from animal models suggests that repeated painful stimuli may result in structural and functional reorganization of the nervous system and alteration in future pain response. Early pain experience during this critical period in development are thought to have immediate and long term consequences that could influence physiological, behavioral and developmental outcomes. Early repetitive procedural pain related stress in very preterm neonates is associated with poorer neurobehaviour in first 2 years of life.1 This study aims to assess the effect of repeated painful stimuli on short term neurobehaviour of preterm infants and the efficacy of repeated doses of sucrose used for pain relief.

DETAILED DESCRIPTION:
DEFINITION OF PAIN - an unpleasant sensory and emotional experience with actual or potential damage or described in terms of such damage (note that the inability to communicate verbally or non verbally does not negate the possibility that an individual is having pain and is in need of appropriate pain relieving treatment)

HISTORICAL BACKGROUND- we as clinicians have emerged from a period of relative neglect of neonatal pain and are now recognizing the immediate and long term impact of pain on the neonatal development as well as the need to alleviate pain effectively. Neonatal pain has been acknowledged and Paediatric societies such as American Academy of Paediatrics and Canadian paediatric society (2000) have adopted specific guidelines on pain relief in neonates .

LONG TERM EFFECTS OF CHRONIC PAIN -Early repeated procedural pain in NICU has been proposed as one of the factors that may contribute to altered development of cognition ,motor function and behaviour in infants and children born preterm.The vulnerability of preterms is well established due to their lower pain threshold ,sensitization from repeated pain and immature systems for maintaining homeostasis .For infants with extremely immature physiological and neurobehavioural systems ,continual adaptation to repeated challenges induces long term alterations in pain sensitivity, might affect generalized stress arousal systems and potentially affect the developing cytotexture of the brain. The physiologic perturbations associated with early prolonged exposure to episodic pain appear to contribute to altering the rapidly developing stress systems .Exposure to painful procedures in early neonatal period affects the long term neurobehavioural outcome.

.

SCALE USED TO ASSESS SHORT TERM NEUROBEHAVIOUR

NAPI (NEUROBEHAVIOURAL ASSESSMENT OF PRETERM INFANT) -The NAPI is appropriate for infants between 32 weeks post conceptional age and term. It assesses the relative maturity of functioning of preterm infants,with higher scores reflecting higher maturity , and can differentiate 2 weeks PCA . The clinical validity and sensitivity of NAPI were established using an index of medical complications based on a 1-5 classification range of degrees of complications21 The items in the motor development cluster include ventral suspension, prone head raising ,the crawling reflex ,forearm recoil ,power of active movements , and vigor of spontaneous movements .The alertness and orientation items include percent of time in an alert state ,duration and quality of alertness , quantitative response to inanimate and animate visual and auditory stimulation and qualitative ratings that express the nature of response.

LACUNAE IN KNOWLEDGE -Preterm infants are more prone to undergo multiple painful procedures due to their prolonged stay in the neonatal intensive care unit and their typical vulnerable clinical profile.It has now been proved that painful procedures lead to long term changes in the pain reactivity and also affect the long term neurobehavioural outcome in these preterm infants.When a medline search was carried out on the subject it did not return any result.Currently there is no study which has tried to explore the short term neurobehavioural outcome in preterm babies >32 weeks - <37 weeks of gestation who undergo multiple painful procedures during their NICU stay.The present study was thus planned to evaluate the role of sucrose analgesia in alleviating the pain caused by the routine NICU procedures over a period of 7 days and to assess the early neurobehavioural outcome in these babies with the help of a well designed double blinded randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. All preterms (more than equal to 32 weeks to less than 37 weeks)
2. within first 48 hrs of post natal life
3. Clinically stable from respiratory and hemodynamic point of view
4. Parental consent

Exclusion Criteria:

1. neonates requiring ventilatory support
2. neonates with any neurological impairment(HIE ,seizures)
3. receiving opiates or born to mothers receiving opiates
4. newborns who have received muscle relaxants ,sedatives or analgesics
5. grade 3 or 4 IVH
6. major congenital anomalies
7. 5 mins apgar of less than 7
8. Neonates undergoing any surgery
9. Birth trauma

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2010-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Short term neurobehaviour status at enrollment in the study and at 40weeks post conceptional age using the NAPI scale. | 40 weeks of post conceptional age.
  Short term neurobehaviour status at enrollment in the study and at 40weeks post conceptional age using the(Neurobehavioural Assessment of Preterm Infant) NAPI scale.

CONTACTS AND LOCATIONS:
Overall Officials: VIKRAM DATTA, MD, Study Chair — Lady Hardinge Medical College
Locations (2):
- India (2):
  - Lady Hardinge Medical College, New Delhi, New Delhi
  - Lady Hardinge Medical College,New Delhi, Delhi